CLINICAL TRIAL: NCT02866591
Title: Interest of Self-compression Technique on Tolerance of Mammography
Acronym: ITACTs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012-A00248-35
Record Dates: First submitted 2016-08-10; First posted 2016-08-15 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: mammography; pain; quality of life; screening; image quality; radiology
MeSH Terms: conditions — Breast Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Patients have a mammography performed by themselves according to auto-compression procedure. The radiologist leads the compression at a minimum threshold of 40 Newton, then leaves the control of the compression to the patient. The radiologist treats only the positioning of the breast on the sensor.
  Interventions: Other: mammography according to an auto-compression procedure; Other: questionary
- Arm B (Active Comparator): Patients have a mammography performed by the radiologist according to standard procedure.
  Interventions: Other: mammography according to a standard procedure; Other: questionary

INTERVENTIONS:
Other: mammography according to an auto-compression procedure
  Arms: Arm A
Other: mammography according to a standard procedure
  Arms: Arm B
Other: questionary

SUMMARY:
Mammography is used for screening, diagnosis, therapeutic evaluation and monitoring of local cancer breast.

It is sometimes poorly tolerated by some patients who complain of an uncomfortable examination or pain.

Breast compression by the manipulator aims to reduce the thickness of the breast during mammography; This act is an important factor of pain or discomfort felt by the patient. But, it is also an image quality factor.

This study aimed to compare self-breast compression by the patient to the compression standard technique carried out by the manipulator.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years and ≤ 75 years of age
* ECOG performance <2
* Mammography planned as part of a breast cancer screening or a monitoring following treatment of a breast lesion
* Ability to provide written informed consent
* Patient's legal capacity to consent to study participation and to understand and comply with the requirements of the study.

Exclusion Criteria:

* Eastern Cooperative Oncology Group performance status ≥ 2
* Treatment for benign lesion with surgery for less than 3 years
* Treatment for cancer with surgery and / or radiotherapy for less than 3 years
* Biopsy for less than 1 year
* Breast prosthesis
* Mastectomy
* Assessment motivated by a clinical breast abnormality

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Comparison of two breast compression techniques (auto-compression versus standard procedure) in mammography | 1 day
  The comparison will be evaluated by the thickness (mm) of breast compressed

SECONDARY OUTCOMES:
Overall tolerance of mammography | 1 day
  The overall tolerance of mammography will be assessed by the patient after 4 shots. The pain felt by the patient will be assessed using a visual analog scale.
Breast compression force | 1 day
  Value measured on compressive force console (Newtons)
Thickness / compressing force ratio | 1 day
Image quality | 1 day
  The image quality will be assessed by the radiologist with a quotation of motion blurring on a 4-point scale
Overall assessment of the manipulator | 1 day
  The appreciation of the manipulator will be assessed using a 4-point scale
Overall assessment of self-satisfaction of the patient at the end of the examination | 1 day
  The measurement of patient satisfaction will be evaluated using a self-administered Norwegian questionnaire (MammoGraphy Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: HENROT Philippe, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (6):
- France (6):
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Cabinet de radiologie, Nancy
  - Polyclinique Majorelle, Nancy
  - Institut Curie, Paris
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henrot P, Boisserie-Lacroix M, Boute V, Troufleau P, Boyer B, Lesanne G, Gillon V, Desandes E, Netter E, Saadate M, Tardivon A, Grentzinger C, Salleron J, Oldrini G. Self-compression Technique vs Standard Compression in Mammography: A Randomized Clinical Trial. JAMA Intern Med. 2019 Mar 1;179(3):407-414. doi: 10.1001/jamainternmed.2018.7169. PMID 30715083